CLINICAL TRIAL: NCT03008213
Title: Fixed Dose Combination of Netupitant and Palonosetron (Akynzeo®) in the Treatment of Refractory Chemotherapy-Induced Nausea and Vomiting
Brief Title: Combination of Netupitant and Palonosetron (Akynzeo®) in the Treatment of Refractory CINV
Acronym: CINV
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI is leaving UCSD
Sponsor: Joseph Ma (Other)
Responsible Party: Sponsor-Investigator, Joseph Ma, Associate Clinical Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UCSD
Record Dates: First submitted 2016-12-14; First posted 2017-01-02 (Estimated); Results first posted 2019-05-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Chemotherapy Induced Nausea Vomiting
MeSH Terms: interventions — netupitant, palosentron drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Netupitant and Palonosetron (Experimental): Subjects will be allowed to participate only once in the study. Study Day 1 will be the day of Akynzeo® dosing. Subjects will receive a single capsule of Akynzeo® (300 mg of netupitant and 0.5 mg of palonosetron) on Study 1.
  Interventions: Drug: Netupitant and Palonosetron

INTERVENTIONS:
Drug: Netupitant and Palonosetron — 300 mg of netupitant and 0.5 mg of palonosetron
  Other Names: Akynzeo

SUMMARY:
Prevention and control of Chemotherapy-Induced Nausea and Vomiting (CINV) are most important in treatment of cancer patients. CINV is one of the most distressing severe side effects of cancer treatment and can have a significant impact on a patient's quality of life. The chemotherapy agents that cause the worst degree of nausea and vomiting are categorized into two groups: moderately emetogenic chemotherapy (MEC) and highly emetogenic chemotherapy (HEC). Nausea and vomiting that occurs within the first day of the administration of chemotherapy agents is considered acute CINV, while nausea and vomiting following 24 hours of the administration of chemotherapy agents is considered delayed CINV. Refractory CINV occurs when patients develop CINV during subsequent cycles of chemotherapy when drugs preventing vomiting and nausea (antiemetic prophylaxis) has not been successful in controlling CINV in earlier cycles. The purpose of this study is to assess the efficacy of Akynzeo in the treatment of refractory CINV

DETAILED DESCRIPTION:
This is a Phase II, single-center, single-arm, open-label, feasibility trial using a fixed dose combination of netupitant and palonosetron (Akynzeo®) in the treatment of refractory CINV. The primary aim of this study is feasibility, defined as 70% completion rate of all study procedures over 7 days.

Eligible subjects will be identified in weekly palliative care patient triage meetings. Patients who are 18 years of age or older, have histologically confirmed cancer, and confirmed refractory CINV will be eligible. After obtaining written informed consent and verifying that the study subject meets all eligibility criteria, the subject will be enrolled in the study through the University California San Diego (UCSD) Moores Cancer Center Clinical Trials Office. Subjects will be allowed to participate only once in the study. Study Day 1 will be the day of Akynzeo® dosing. Subjects will receive a single capsule of Akynzeo® (300 mg of netupitant and 0.5 mg of palonosetron) on Study 1. Study drug may be taken with or without food. Subjects will complete a study drug diary to document date and time of Akynzeo® administration. On Study Day 1, the study coordinator will educate the subject on how to complete the Multinational Association of Supportive Care in Cancer (MASCC) Antiemesis Tool, and Functional Living Index Emesis (FLIE) scale, and medication diary and each of these documents will be completed for that day. An adequate number of copies of each subject questionnaire and diary will be provided to the subject on Study Day 1 for completion at home during the post-treatment observation portion of the study (Study Days 2-7) as needed.

ELIGIBILITY:
Inclusion Criteria:

1. Adults greater than or equal to 18 years old.
2. Must have a histologically confirmed cancer diagnosis.
3. Must have refractory CINV defined as nausea and/or vomiting that occurs after the first cycle of chemotherapy despite guideline-based prophylaxis and after first-line rescue medication with either a dopamine receptor antagonist, steroid, and/or benzodiazepine.
4. Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
5. Life expectancy greater than 3 months.
6. Corrected serum calcium level less than or equal to 10.5 mg/dL.
7. Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 14 days following completion of therapy.

   A) A woman of child-bearing potential is any female (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

   i) Has not undergone a hysterectomy or bilateral oophorectomy; or ii) Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has not had menses at any time in the preceding 12 consecutive months)
8. Women of child-bearing potential must have a negative pregnancy test prior to initiating study treatment.
9. Ability to understand and willingness to sign a written informed consent.

Exclusion Criteria:

1. Patients with QTc interval greater than 450 ms.
2. Patients with a known hypersensitivity reaction to 5-HT3 receptor antagonists or NK1 receptor antagonists.
3. Patients who have taken any medication classified as a strong CYP3A4 inducer within one week of Study Day 1 or 5 halflives (whichever is longer) or use of a strong or moderate CYP3A4 inhibitor within one week of Study Day 1 or 5 halflives (whichever is longer) (see Appendix 2).
4. Patients with severe hepatic impairment as defined as AST/ALT greater than three times the upper limit of normal, total bilirubin greater than 3 mg/dL, and/or Child-Pugh score >9.
5. Patients with end-stage renal disease defined as creatinine clearance of <15mL/min and/or diagnosed with Stage 5 chronic kidney disease.
6. Pregnant or lactating females are excluded from enrollment on this trial.
7. Patients unable to swallow oral medications. Any other condition that, in the opinion of the investigator, may impact the absorption of oral medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-01; Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Ma, PharmD, Principal Investigator — UCSD

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Netupitant and Palonosetron
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Netupitant and Palonosetron
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Completed All Study Procedures Over Seven Days
Description: The proposed study is a prospective, single-center, feasibility trial. The primary aim of this study is feasibility - specifically feasibility will be defined as completion of all study procedures over seven days.
  For the primary aim, we assume an acceptable completion rate from strata of MEC/HEC or tumor types of all study-related procedures would be at least 70%. Assuming a true completion rate of 85%, a sample size of 50 patients would have an 80% power to detect an absolute difference of 15% at Type I error 0.05.
Time Frame: Through study completion, 7 days
Measure: Number; unit: participants
Arm/Group | Netupitant and Palonosetron
Number analyzed (Participants) | 1
participants | 1

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Netupitant and Palonosetron
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Netupitant and Palonosetron (N=1)
nausea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-04): https://cdn.clinicaltrials.gov/large-docs/13/NCT03008213/Prot_SAP_000.pdf